CLINICAL TRIAL: NCT02745951
Title: HELIox CardiOPlegia Trial During Cardiac surgERy
Acronym: HELICOPTER-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15 - 311
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: cardiopulmonary bypass; cardioplegia; cardioprotection; coronary artery bypass graft surgery; heliox
MeSH Terms: interventions — heliox; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heliox (Experimental): Cardioplegia enriched with a 70:30 (Helium:Oxygen) Heliox mixture while the patient is on cardiopulmonary bypass
  Interventions: Other: Heliox
- Standard of care (Active Comparator): Cardioplegia enriched with a Nitrogen and Oxygen mixture while the patient is on cardiopulmonary bypass
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Heliox — Half of the study population will be randomly assigned to receive cardioplegia enriched with a 70:30 (Helium:Oxygen) via a D100 pediatric oxygenator. The Heliox itself will need to be administered via an oxygen regulator using a low flowmeter.
  Arms: Heliox
Other: Standard of care — The other half will be randomized to Nitrogen:Oxygen mixture. This will be done through the standard of care cardioplegia apparatus. There will be no novel interventions administered in this group.
  Arms: Standard of care

SUMMARY:
The HELICOPTER-1 Trial is a single centre pilot study to determine the feasibility of administering Heliox in cardioplegia during cardiac surgery and whether it has the potential to reduce the incidence and severity of myocardial ischemia during and after cardiac surgery.

DETAILED DESCRIPTION:
The HELICOPTER-1 Trial is a single centre, randomized trial evaluating the feasibility of administration of Heliox for prevention of myocardial ischemia in patients undergoing cardiac surgery. Half of the study population will be randomly assigned to the receive cardioplegia enriched with a 70:30 (Helium:Oxygen) Heliox mixture, while the other half will be randomized to receive the current clinical standard of care (nitrogen and oxygen in cardioplegia).

Subjects will be followed up daily during their post-operative course in hospital for clinical outcomes. A 30-day phone follow-up will be conducted for vital status and MI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Cardiac surgery with CPB where use of a coronary sinus catheter is indicated

Exclusion Criteria:

* Patient refusal
* Recent myocardial infarction (less than 7 days old)
* Left ventricular ejection fraction less than 30%
* Known pregnancy on date of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using Heliox to oxygenate the blood cardioplegia | 30 days from the intervention
  To determine the feasibility of using Heliox to oxygenate the blood cardioplegia. Feasibility will be measured according to subject enrollment rates and to measurement of the blood gas content of the cardioplegia solutions.

SECONDARY OUTCOMES:
New Myocardial Infarction | 30 days from the intervention
  Myocardial infarction (MI) will be defined according to the Third Universal Definition of MI using the following two criteria:
  1. Serum levels of Troponin I: Values more than 10 times the 99th percentile of the upper limit from a normal baseline. If preoperative enzyme levels are abnormal, the post-operative enzymes must be greater than the baseline plus 10 times the upper limit from a normal baseline.
  2. ECG: At least one of the following i) New left bundle branch block ii) Development of new pathological Q waves iii) Imaging evidence of new loss of viable myocardium or new regional wall abnormality

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided